CLINICAL TRIAL: NCT02112877
Title: VIRTUS Safety and Efficacy of the Veniti Vici™ Venous Stent System (Veniti, Inc.) When Used to Treat Clinically Significant Chronic Non-malignant Obstruction of the Iliofemoral Venous Segment
Brief Title: VIRTUS: An Evaluation of the Vici™ Venous Stent System in Patients With Chronic Iliofemoral Venous Outflow Obstruction
Acronym: VIRTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STE-HUM-004P; STE-HUM-007P (Other: Sponsor)
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Chronic Venous Disorder; Venous Outflow Obstruction; Symptomatic Venous Outflow Obstruction of Iliofemoral Vein
Keywords: iliofemoral vein; venous; venous obstruction

STUDY DESIGN:
Intervention Model Description: Thirty (30) patients will be enrolled at approximately 7 centers (feasibility cohort). These patients will not be included in the pivotal study population, but will be evaluated separately for the primary safety and efficacy endpoints as well as for all secondary endpoints. When these 30 feasibility patients have completed their 30-day follow-up, a Data Safety Monitoring Board (DSMB) will review the safety data and will determine if the study can proceed with enrollment of the 170 pivotal subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- VICI Stent Implantation - Feasibility (Experimental): Percutaneous stent placement in the common femoral vein, external iliac vein and/or common iliac vein Veniti Vici™ Venous Stent System
  Interventions: Device: Veniti Vici™ Venous Stent System
- VICI Stent Implantation - Pivotal (Experimental): Percutaneous stent placement in the common femoral vein, external iliac vein and/or common iliac vein Veniti Vici™ Venous Stent System
  Interventions: Device: Veniti Vici™ Venous Stent System

INTERVENTIONS:
Device: Veniti Vici™ Venous Stent System

SUMMARY:
This is a prospective, multi-center, single arm, non-randomized study to define safety and efficacy of the Veniti Vici™ Venous Stent System in relation to pre-defined Objective Performance goals. A maximum of 200 patients at up to 45 centers worldwide will be enrolled. Thirty (30) feasibility patients will be enrolled at approximately 7-10 centers and 170 pivotal patients will be enrolled at approximately 45 centers worldwide. The follow-up period is 36 months.

DETAILED DESCRIPTION:
The objective of this prospective study is to assess the safety and efficacy of the Veniti Vici™ Venous Stent System in achieving patency of the target venous lesion in patients who present with clinically significant chronic non-malignant obstruction of the iliofemoral venous outflow tract.

ELIGIBILITY:
Inclusion Criteria - Pre-Procedure Criteria:

* Age ≥ 18 years
* Willing and capable of complying with all follow-up evaluations at the specified times
* Able and willing to provide written informed consent prior to study-specific procedures
* Presence of unilateral, clinically significant, chronic non-malignant obstruction of the common femoral vein, external iliac vein, common iliac vein, or any combination thereof, defined as a ≥50% reduction in target vessel lumen diameter (to be measured by venogram during procedure)
* Clinically significant venous obstruction defined as meeting at least one of the following clinical indicators:

  * Clinical severity class of CEAP classification ≥3
  * VCSS Pain Score ≥2
* Negative pregnancy test in females of child-bearing potential
* Intention to stent the target lesion only with the Veniti Vici Venous Stent

Exclusion Criteria - Pre-Procedure Criteria:

* Presence or history of clinically significant pulmonary emboli within 6 months prior to enrollment.
* Venous obstruction that extends into the inferior vena cava (IVC)
* Contralateral disease of the common femoral vein, external iliac vein, common iliac vein, or any combination thereof with planned treatment within 30 days after subject enrollment
* Life expectancy <12 months
* Female of childbearing potential who is pregnant or plans to become pregnant during the duration of the clinical study
* Uncontrolled or active coagulopathy OR known, uncorrectable bleeding diathesis with the following definitions:

  * Uncorrected INR ≥2.0 or aPTT ≥1.5 X normal local lab value
  * Platelet count <80,000
* Uncorrected hemoglobin of ≤ 9 g/dL
* Patients with an estimated glomerular filtration rate (eGFR) <30 mL/min. In patients with diabetes mellitus, eGFR <45 mL/min.
* Known hypersensitivity to nickel or titanium
* Contrast agent allergy that cannot be managed adequately with pre-medication
* Intended concurrent thrombolysis or thrombectomy procedure OR intended or planned (within 30 days) adjuvant procedure such as creation of temporary arteriovenous fistula, placement of IVC filter, endovenectomy or saphenous vein ablation
* Current or recent (within 30 days) active participation in another drug or device clinical trial (Participation in observational studies is acceptable.)
* Patient judged to be a poor candidate by the primary investigator
* Patients who have had any prior surgical or endovascular intervention of the target vessel [Note: Patients who have had catheter-directed or mechanical thrombolysis in the target vessel for DVT at least 3 month (90 days) prior to the VIRTUS index procedure may be included in the trial.]

Exclusion Criteria - Intra-Procedural Criteria:

* Patients in whom the lesions cannot be traversed with a guide wire.
* Patients where the obstruction extends into the inferior vena cava or below the level of the lesser trochanter.
* Patients whose vein diameters are not within limits stated in current Instructions for Use as determined by venogram.
* Patients who do not meet the venogram binary stenosis definition, as determined by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Marston, MD, Principal Investigator — UNC Department of Surgery; Mahmood Razavi, MD, Principal Investigator — Vascular and Interventional Specialists of Orange County
Locations (24):
- United States (16):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Healthfinity PLCC, Scottsdale, Arizona
  - Arkansas Site Management Services, LLC, Little Rock, Arkansas
  - St. Joseph Hospital, Orange, California
  - Radiology Imaging Associates, Englewood, Colorado
  - Vascular Breakthroughs, Darien, Connecticut
  - Midwest Cardiovascular Foundation, Davenport, Iowa
  - Imperial Health, LLP, Lake Charles, Louisiana
  - Michigan Vascular Center, Flint, Michigan
  - NYU School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Dr. Ediberto Soto-Cora, El Paso, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
- France (2):
  - Infermerierie Protestante de Lyon, Décines-Charpieu
  - Hôpital Nord de Marseille, Marsaille
- Klinikum Arnsberg, Karolinen Hospital, Arnsberg, Germany
- University Hospital Galway, Galway, Ireland
- Rijnstate Ziekenhuis, Arnhem, Netherlands
- University Hospital HM Monteprincipe, Madrid, Spain
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University College London, London

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829
- [Derived] Razavi MK, Black S, Gagne P, Chiacchierini R, Nicolini P, Marston W; VIRTUS Investigators. Pivotal Study of Endovenous Stent Placement for Symptomatic Iliofemoral Venous Obstruction. Circ Cardiovasc Interv. 2019 Dec;12(12):e008268. doi: 10.1161/CIRCINTERVENTIONS.119.008268. Epub 2019 Dec 13. PMID 31833414
- [Derived] Razavi M, Marston W, Black S, Bentley D, Neglen P. The initial report on 1-year outcomes of the feasibility study of the VENITI VICI VENOUS STENT in symptomatic iliofemoral venous obstruction. J Vasc Surg Venous Lymphat Disord. 2018 Mar;6(2):192-200. doi: 10.1016/j.jvsv.2017.10.014. Epub 2017 Dec 28. PMID 29290601

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 200 subjects have been enrolled in the VIRTUS Trial, including 30 subjects in the feasibility cohort and 170 subjects in the pivotal cohort.
Period: Overall Study
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Started | 30 | 170
Completed | 28 | 157
Not Completed | 2 | 13
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Visit Missed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal | Total
Number analyzed (Participants) | 30 | 170 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (14.3) | 54.4 (16.2) | 52.9 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 96 | 120
  Male | 6 | 74 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 5 | 7
  Black or African American | 1 | 20 | 21
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  White | 25 | 127 | 152
  White African | 0 | 1 | 1
  Latin American | 0 | 1 | 1
  Not Answered | 0 | 14 | 14
  North African | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: For the feasibility cohort, ethnicity data has been provided by 27/30 subjects. For the pivotal cohort, 16 subjects from the sites located in France did not provide their ethnicity per the policy at each site.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 27 | 154 | 181
    Hispanic or Latino | 2 | 13 | 15
    Not Hispanic or Latino: number analyzed (Participants) | 27 | 154 | 181
    Not Hispanic or Latino | 25 | 141 | 166
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 1 | 0 | 1
  United States | 8 | 119 | 127
  Ireland | 3 | 5 | 8
  United Kingdom | 10 | 22 | 32
  France | 3 | 18 | 21
  Germany | 0 | 5 | 5
  Spain | 5 | 1 | 6
Chronic Non-Malignant Obstruction [Count of Participants; unit: Participants]
  Left Leg | 24 | 145 | 169
  Right Leg | 5 | 24 | 29
  Both Legs | 1 | 1 | 2
Clinical Etiology Anatomy Pathophysiology (CEAP) Assessment [Count of Participants; unit: Participants]
  0 (No visible or palpable signs of venous disease | 1 | 2 | 3
  1 (Telangiectasia or reticular veins) | 0 | 0 | 0
  2 (Varicose Veins) | 0 | 2 | 2
  3 (Edema) | 13 | 45 | 58
  4 (Skin changes ascribed to venous disease) | 13 | 78 | 91
  5 (Healed ulceration) | 2 | 22 | 24
  6 (Active ulceration) | 1 | 21 | 22
Venous Clinical Severity Score (VCSS) Leg Pain (Target Limb) [Count of Participants; unit: Participants] — Population: For the pivotal cohort, results for 24 subjects from a single US center are not included due to data integrity issues.
  Participants
    Absent: number analyzed (Participants) | 30 | 146 | 176
    Absent | 2 | 15 | 17
    Mild: number analyzed (Participants) | 30 | 146 | 176
    Mild | 2 | 35 | 37
    Moderate: number analyzed (Participants) | 30 | 146 | 176
    Moderate | 17 | 54 | 71
    Severe: number analyzed (Participants) | 30 | 146 | 176
    Severe | 9 | 42 | 51
Diabetic [Count of Participants; unit: Participants] | 2 | 29 | 31
Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 3 | 21 | 24
  Former Smoker | 8 | 41 | 49
  Non-Smoker | 19 | 108 | 127
History of Pulmonary Embolism (PE) [Count of Participants; unit: Participants] — Population: For the feasibility cohort, only 19 subjects were initially classified as having a history of thromboembolic disease. For the pivotal cohort, only 130 subjects were initially classified as having a history of thromboembolic disease.
  Participants
    number analyzed (Participants) | 19 | 130 | 149
    (all) | 2 | 28 | 30
History of Deep Vein Thrombosis (DVT) [Count of Participants; unit: Participants] — Population: For the feasibility cohort, only 19 subjects were initially classified as having a history of thromboembolic disease. For the pivotal cohort, only 130 subjects were initially classified as having a history of thromboembolic disease.
  Participants
    number analyzed (Participants) | 19 | 130 | 149
    (all) | 19 | 119 | 138
History of Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 0 | 14 | 14
History of Myocardial Infarction (MI) within past 5 years [Count of Participants; unit: Participants] | 0 | 1 | 1
History of Coronary Artery Bypass Grafting (CABG) [Count of Participants; unit: Participants] | 0 | 4 | 4
History of Percutaneous Transluminal Coronary Angioplasty (PTCA)/Stent [Count of Participants; unit: Participants] | 0 | 4 | 4
History of Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] | 0 | 4 | 4
History of Hypertension (HTN) [Count of Participants; unit: Participants] | 7 | 68 | 75
History of Hepatic Disease [Count of Participants; unit: Participants] | 1 | 5 | 6
History of Renal Disease [Count of Participants; unit: Participants] | 1 | 8 | 9
History of Peripheral Vascular Disease (PVD) [Count of Participants; unit: Participants] | 2 | 29 | 31
History of Coagulation Disorder [Count of Participants; unit: Participants] | 7 | 23 | 30
History of Cerebrovascular Accident (CVA) [Count of Participants; unit: Participants] | 1 | 10 | 11
History of Cancer [Count of Participants; unit: Participants] | 2 | 18 | 20
History of Recent Trauma [Count of Participants; unit: Participants] | 1 | 3 | 4
History of Allergies [Count of Participants; unit: Participants] | 4 | 60 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: The primary safety endpoint for this study will be a composite endpoint of any major adverse event (MAE) within 30 days, as adjudicated by a Clinical Events Committee.
Time Frame: 30 days
Population: For the pivotal cohort, one subject never returned for follow-up after discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 30 | 169
Participants
  Device or procedure-related death | 0 | 0
  Device or procedure-related bleeding | 0 | 0
  Device or procedure-related arterial/venous injury | 2 | 2
  Device or procedure-related acuteDeepVeinThrombus | 0 | 0
  Clinically significant pulmonary embolism | 0 | 0
  Embolization of the stent | 0 | 0

2. Primary Outcome: Percentage of Participants That Demonstrated Primary Patency
Description: The primary effectiveness endpoint is the primary patency rate at 12 months post-intervention, defined as freedom from occlusion by thrombosis, freedom from surgical or endovascular intervention on target vessel which are found to have re-stenosis or stent occlusion to maintain patency, and freedom from in-stent stenosis more than 50% by venogram.
Time Frame: 12 months post-intervention
Population: For the feasibility cohort, month 12 outcomes were available for 22 subjects. For the pivotal cohort, month 12 outcomes were available for 125 subjects. Those without venography performed at 12 months had their result assigned by random selection from subjects with a venogram result who had the same anatomy and the same DUS outcome (if available).
Measure: Number; unit: Percentage of Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 22 | 170
Percentage of Participants | 77.3 | 84.0

3. Secondary Outcome: Number of Participants With Improvement in Venous Clinical Severity Score (VCSS)
Description: The secondary effectiveness endpoint for this study will be a binary response variable based on an improvement in Venous Clinical Severity Score (VCSS) by at least 50% at 12 months post-intervention. VCSS measures 10 clinical attributes of venous disease (Pain, Varicose Veins, Venous Edema, Skin Pigmentation, Inflammation, Induration, No. Active Ulcers, Active Ulcer Size, Ulcer Duration and Compression Therapy) on a scale of 0 - 3 (Absent 0, Mild 1, Moderate 2, and Severe 3).
Time Frame: 12 months post-intervention
Population: For the feasibility cohort, 7 subjects did not have VCSS results at both month 12 and baseline. For the pivotal cohort, results for 24 subjects from a single US center are not included due to data integrity issues and 14 subjects did not have VCSS results at both month 12 and Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 23 | 132
Participants | 13 | 65

4. Other Pre Specified Outcome: Number of Participants With Procedural Technical Success
Description: Procedural technical success is achievement of a final residual target vessel diameter stenosis of ≤50% as measured on the post procedural venogram, without skipped lesion regions, with placement of the study device alone with or without post-stenting balloon dilation as needed.
Time Frame: During Procedure
Population: For the pivotal cohort, four subjects did not have the post-procedural venogram available for assessment. Additionally, there were two subjects that failed the endpoint due to two investigators using non-study stents.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 30 | 166
Participants | 30 | 164

5. Other Pre Specified Outcome: Number of Participants With Lesion Success
Description: Lesion success is defined as achievement of ≤50% residual diameter stenosis of the target lesion using any percutaneous method (including the use of non-study devices).
Time Frame: During Procedure
Population: For the pivotal cohort, four subjects did not have the post-procedural veogram available for assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 30 | 166
Participants | 30 | 166

6. Other Pre Specified Outcome: Number of Participants With Procedural Success
Description: Procedural success is defined as procedural technical success without the occurrence of a major adverse event (MAE) between the index procedure and discharge.
Time Frame: From the time of the Index Procedure post procedural venogram through the time of Index Procedure Discharge or 3 days Post-Procedure (whichever comes first)
Population: For the pivotal cohort, four subjects did not have the post-procedural venogram available for assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 30 | 166
Participants | 28 | 162

7. Other Pre Specified Outcome: Number of Participants With Late Technical Success
Description: Late technical success (through 12 months) is the absence of device movement >10mm related to anatomical landmarks or any migration leading to symptoms or requiring therapy; absence of stent occlusion by thrombosis or restenosis, defined as reduction in treated segment lumen more than 50% from the post-procedure vessel lumen diameter as measured by post-procedural venogram or DUS and maintenance of structural integrity, defined as the absence of pinching (focal compression), kinking (stent doubling or bending upon itself) that results in >50% diameter reduction of the stent, recoil (poor radial resistive force) or absence of fractures .
Time Frame: 12 months post-intervention
Population: For the feasibility cohort, month 12 outcomes were available for 22 subjects. For the pivotal cohort, only 127 subjects had a 12-month venogram and/or stent fracture assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 22 | 127
Participants | 16 | 97

8. Other Pre Specified Outcome: Change in the Quality of Life (Chronic Venous Insufficiency Questionnaire)(CIVIQ2))
Description: The overall change in CIVIQ2 scores for the study patients, calculated using the mean scores at baseline and 12-months. This instrument is scored from 20 to 100 points with lower scores indicating a lesser impact on health.
Time Frame: Baseline and 12 months post-intervention
Population: For the feasibility cohort, three subjects did not have Month 12 CIVIQ-2 results. For the pivotal cohort, results for 24 subjects from a single US center are not included due to data integrity issues. Also, 11 subjects did not have a Month 12 visit and 2 subjects did not complete the CIVIQ forms.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 27 | 133
units on a scale | -15.4 [-22.1 to -8.6] | -13.1 [-16.3 to -10.0]

9. Other Pre Specified Outcome: Number of Participants With Estimated Primary-Assisted Patency
Description: Primary-assisted patency is defined as freedom from occlusion regardless of whether an intervention (subsequent to the index procedure) was performed.
Time Frame: 12 months post-intervention
Population: For the feasibility cohort, only 21 subjects had known outcomes. For the pivotal cohort, only 126 subjects had known outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 21 | 126
Participants | 20 | 117

10. Other Pre Specified Outcome: Number of Participants With Estimated Secondary Patency
Description: Secondary patency is defined as freedom from "permanent" loss of patency determined through last follow-up (irrespective of the number of interventions).
Time Frame: 36 months post-intervention
Population: For the feasibility cohort, 13 subjects had known outcomes. For the pivotal cohort, 97 subjects had known outcomes.
Measure: Count of Participants; unit: Participants
Groups:
- VICI Stent Implantation - Feasibility; VICI Stent Implantation - Pivotal: Percutaneous stent placement in the common femoral vein, external iliac vein and/or common iliac vein Veniti Vici™ Venous Stent System
  Veniti Vici™ Venous Stent System
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
Number analyzed (Participants) | 13 | 97
Participants | 13 | 93

ADVERSE EVENTS:
Time Frame: Adverse event data were collected to one year post-implant, up to 12 months. Serious adverse event data were collected to one year post-implant, and will be collected up to 60 months.
Arm/Group | VICI Stent Implantation - Feasibility | VICI Stent Implantation - Pivotal
All-Cause Mortality (participants affected / at risk) | 0/30 | 4/170
Serious Adverse Events (participants affected / at risk) | 14/30 | 86/170
Other Adverse Events (participants affected / at risk) | 14/30 | 102/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VICI Stent Implantation - Feasibility (N=30) | VICI Stent Implantation - Pivotal (N=170)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 4 (6) | 10 (14)
Vascular stent restenosis (General disorders) | 2 (2) | 8 (9)
Vascular stent stenosis (General disorders) | 2 (3) | 4 (5)
Vascular stent occlusion (General disorders) | 1 (1) | 2 (2)
Stenosis (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 3 (4)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular access site hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalized ratio decreased (Investigations) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3)
Specific gravity urine abnormal (Investigations) | 0 (0) | 1 (1)
Renal vein compression (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Venous angioplasty (Surgical and medical procedures) | 4 (7) | 9 (11)
Venous stent insertion (Surgical and medical procedures) | 3 (3) | 2 (2)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Thrombolysis (Surgical and medical procedures) | 0 (0) | 4 (4)
Vascular stent insertion (Surgical and medical procedures) | 0 (0) | 2 (2)
Angioplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Thrombectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Varicose vein operation (Surgical and medical procedures) | 2 (2) | 4 (4)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Myomectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Transfusion (Surgical and medical procedures) | 0 (0) | 2 (2)
Interventional procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 2 (2)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 17 (24)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 2 (3)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Varicose ulceration (Vascular disorders) | 0 (0) | 1 (1)
Vascular compression (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (2)
Stent malfunction (Product Issues) | 2 (2) | 2 (2)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 0 (0) | 6 (15)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4)
Cellulitis (Infections and infestations) | 0 (0) | 8 (11)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Paget-Schroetter syndrome (Vascular disorders) | 0 (0) | 1 (1)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheterisation venous (Surgical and medical procedures) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 3 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Atherectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Neurolysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (2)
Anal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thecal sac compression (Nervous system disorders) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pelvic congestion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergy to plants (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VICI Stent Implantation - Feasibility (N=30) | VICI Stent Implantation - Pivotal (N=170)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhaea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile acid malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Tenderness (General disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1) | 5 (5)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 16 (17)
Chest pain (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Vascular stent occlusion (General disorders) | 0 (0) | 3 (3)
Puncture site hemorrhage (General disorders) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 0 (0) | 2 (2)
Localized oedema (General disorders) | 0 (0) | 1 (1)
Vascular stent restenosis (General disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Infected varicose vein (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Root canal infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1)
Antiphospholipid antibodies positive (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 (0) | 1 (1)
Venous pressure increased (Investigations) | 0 (0) | 1 (1)
Cyst aspiration (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 15 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 17 (21)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnaea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Venous angioplasty (Surgical and medical procedures) | 0 (0) | 3 (3)
Thrombolysis (Surgical and medical procedures) | 0 (0) | 2 (2)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Joint fluid drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Vena cava filter insertion (Surgical and medical procedures) | 0 (0) | 1 (2)
Vena cava filter removal (Surgical and medical procedures) | 0 (0) | 1 (2)
Vascular stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Venous stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Hyperemia (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 16 (25)
Phlebitis (Vascular disorders) | 0 (0) | 2 (2)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Surgical and medical procedures) | 0 (0) | 2 (2)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Varicose ulceration (Vascular disorders) | 0 (0) | 1 (2)
Vascular insufficiency (Vascular disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Phonophobia (Psychiatric disorders) | 0 (0) | 1 (1)
Drug use disorder (Psychiatric disorders) | 0 (0) | 2 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic congestion (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Homeless (Social circumstances) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Stent malfunction (Product Issues) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT02112877/Prot_SAP_000.pdf